CLINICAL TRIAL: NCT01196000
Title: Laparoscopic Versus Robotic-Assisted Surgery for Rectal Cancer
Brief Title: Laparoscopic Surgery or Robotic-Assisted Laparoscopic Surgery in Treating Patients With Rectal Cancer That Can Be Removed By Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has never been opened to accrual at COH. Study to be closed at COH due to the lack of qualified robotic colorectal surgeons.
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07158; NCI-2010-01427
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Recurrent Rectal Cancer; Stage I Rectal Cancer; Stage II Rectal Cancer; Stage III Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients undergo standard conventional laparoscopic resection.
  Interventions: Procedure: conventional laparoscopic surgery; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm II (Experimental): Patients undergo robotic-assisted laparoscopic resection.
  Interventions: Procedure: robotic-assisted laparoscopic surgery; Procedure: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Procedure: conventional laparoscopic surgery — operation using conventional laparoscopic techniques
  Other Names: laparoscopy-assisted surgery; surgery, laparoscopic
  Arms: Arm I
Procedure: robotic-assisted laparoscopic surgery — operation that involves use of laparoscopic assistance with robotic assistance
  Arms: Arm II
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
RATIONALE: Robotic-assisted laparoscopic surgery may be a less invasive type of surgery for rectal cancer and may have fewer side effects and improve recovery. It is not yet known whether robotic-assisted laparoscopic surgery is more effective than laparoscopic surgery in treating patients with rectal cancer.

PURPOSE: This randomized clinical trial studies robotic-assisted laparoscopic surgery to see how well it works compared to laparoscopic surgery in treating patients with rectal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To evaluate robotic-assisted rectal cancer surgery versus standard laparoscopic rectal cancer resection by means of a randomized, controlled trial.

II. To assess technical ease of the operation, as determined by the clinical indicator of low conversion rate to open operation.

III. To assess surgical accuracy and improved oncological outcome as determined by clear pathological resection margins.

IV. To assess quality of life and analyze cost-effectiveness to aid evidence-based knowledge to inform NHS and other service providers and decision-makers.

V. To analyze disease-free and overall survival and local recurrence rates at 3-year follow-up.

OUTLINE:

Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo standard laparoscopic resection.

ARM II: Patients undergo robotic-assisted laparoscopic resection.

After completion of study treatment, patients are followed up at 1 month, 6 months, and then annually thereafter for 3 years.

ELIGIBILITY:
Inclusion

* Able to provide written informed consent
* Diagnosis of rectal cancer amenable to curative surgery either by anterior resection or abdominoperineal resection (i.e. staged T1-3, N0-2, M0 by CT and MRI or transrectal ultrasound)
* Rectal cancer suitable for resection by either standard or robotic-assisted laparoscopic procedure
* Fit for robotic-assisted or standard laparoscopic rectal resection
* ASA =< 3
* Capable of completing required questionnaires at time of consent

Exclusion

* Benign lesions of the rectum
* Cancers of the anal canal
* Locally advanced cancers not amenable to curative surgery
* Locally advanced cancers requiring en bloc multi-visceral resection
* Synchronous colorectal tumours requiring multi-segment surgical resection
* Co-existent inflammatory bowel disease
* Clinical or radiological evidence of metastatic spread
* Concurrent or previous diagnosis of invasive cancer within 5 years that could confuse diagnosis (non-melanomatous skin cancer or superficial bladder cancer treated with curative intent are acceptable; for other cases please discuss with Chief Investigator via CTRU)
* History of psychiatric or addictive disorder or other medical condition that, in the opinion of the investigator, would preclude the patient from meeting the trial requirements
* Pregnancy
* Participation in another rectal cancer clinical trial relating to surgical technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Rate of conversion to open surgery as an indicator of surgical technical difficulty | At completion of surgery

SECONDARY OUTCOMES:
Circumferential resection margin positivity rate | At completion of pathology review
Local recurrence rate | At 3 years
Intra-operative and post-operative complications | At day 30 and 6 months
Operative mortality | At day 30
Self reported bladder and sexual function | At day 30 and 6 months
Health related quality of life | At day 30 and 6 months
Disease free and overall survival | At 3 years
Intra-operative laparoscopic skills (randomly selected cases only) as assessed by the global assessment tool for evaluation of intra-operative laparoscopic skills (GOALS) | Upon completion of GOALS assessment by an independent expert
Quality of the plane of surgery as assessed by central review of photographs | At completion of the central review of photographs
Health economics | At day 30 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Pigazzi, Principal Investigator — City of Hope Medical Center